CLINICAL TRIAL: NCT04416932
Title: Advanced Imaging for Shoulder and Elbow Arthroplasty
Brief Title: Ultrasound After Total Shoulder Arthroplasty
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Piedmont Orthopedic Society (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00103782
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Total Shoulder Arthroplasty; Rotator Cuff Tears; Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-operative patients who had total shoulder arthroplasty: Patients who have had a total shoulder replacement will be scheduled for an ultrasound at Duke Radiology. An ultrasound will be completed on the shoulder that has been replaced, which takes no more than an hour. This ends all study involvement.
  Interventions: Procedure: Ultasound

INTERVENTIONS:
Procedure: Ultasound — Evaluation of post-operative patients who have had total shoulder arthroplasty and will assess the integrity of the rotator cuff using ultrasound.

SUMMARY:
The purpose of this study would be to evaluate a group of patients status post post-total shoulder arthroplasty to assess the integrity of the rotator cuff using ultrasound. We believe ultrasonography imaging to be a comparable and efficacious modality to evalute tenotomy healing rates and diagnose rotator cuff failure after total shoulder arthroplasty. In addition, we believe ultrasonography to be a cost-effective modality to asses the rotator cuff after total shoulder arthroplasty. Our population would consist of patients that received total shoulder arthroplasty within the last 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Primary or revision total shoulder arthroplasty with or without subscapularis tenotomy
* Primary or revision reverse shoulder arthroplasty with or without subscapularis tenotomy
* English speaking patients only
* Shoulder arthroplasty within the last 5 years

Exclusion Criteria:

* Revision shoulder arthroplasty for infection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Duke patients who have had prior total shoulder arthroplasy surgery within the past 5 years who are 18 years of age or older.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Number of confirmed healed rotator cuff tear as measured by ultrasound | time of procedure, up to 1 hour
Number of confirmed non-healed tenotomy | time of procedure, up to 1 hour
Number of confirmed rotator cuff tears | time of procedure, up to 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Klifto, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong A, Lashgari C, Teefey S, Menendez J, Yamaguchi K, Galatz LM. Ultrasound evaluation and clinical correlation of subscapularis repair after total shoulder arthroplasty. J Shoulder Elbow Surg. 2006 Sep-Oct;15(5):541-8. doi: 10.1016/j.jse.2005.09.013. Epub 2006 Jul 27. PMID 16979047
- [Background] Dines JS. Editorial Commentary: Rotator Cuff Surgery Planning: Yet Another Reason for Orthopedic Surgeons to Learn to Use Ultrasound.... Arthroscopy. 2018 Aug;34(8):2285-2286. doi: 10.1016/j.arthro.2018.06.019. PMID 30077254
- [Background] Gilat R, Atoun E, Cohen O, Tsvieli O, Rath E, Lakstein D, Levy O. Recurrent rotator cuff tear: is ultrasound imaging reliable? J Shoulder Elbow Surg. 2018 Jul;27(7):1263-1267. doi: 10.1016/j.jse.2017.12.017. Epub 2018 Feb 3. PMID 29398398
- [Background] Horner NS, de Sa D, Heaven S, Simunovic N, Bedi A, Athwal GS, Ayeni OR. Indications and outcomes of shoulder arthroscopy after shoulder arthroplasty. J Shoulder Elbow Surg. 2016 Mar;25(3):510-8. doi: 10.1016/j.jse.2015.09.013. Epub 2015 Dec 2. PMID 26652703
- [Background] Iannotti JP, Ciccone J, Buss DD, Visotsky JL, Mascha E, Cotman K, Rawool NM. Accuracy of office-based ultrasonography of the shoulder for the diagnosis of rotator cuff tears. J Bone Joint Surg Am. 2005 Jun;87(6):1305-11. doi: 10.2106/JBJS.D.02100. PMID 15930541
- [Background] Karthikeyan S, Rai SB, Parsons H, Drew S, Smith CD, Griffin DR. Ultrasound dimensions of the rotator cuff in young healthy adults. J Shoulder Elbow Surg. 2014 Aug;23(8):1107-12. doi: 10.1016/j.jse.2013.11.012. Epub 2014 Jan 16. PMID 24439247
- [Background] Levy DM, Abrams GD, Harris JD, Bach BR Jr, Nicholson GP, Romeo AA. Rotator cuff tears after total shoulder arthroplasty in primary osteoarthritis: A systematic review. Int J Shoulder Surg. 2016 Apr-Jun;10(2):78-84. doi: 10.4103/0973-6042.180720. PMID 27186060
- [Background] Narasimhan R, Shamse K, Nash C, Dhingra D, Kennedy S. Prevalence of subscapularis tears and accuracy of shoulder ultrasound in pre-operative diagnosis. Int Orthop. 2016 May;40(5):975-9. doi: 10.1007/s00264-015-3043-9. Epub 2015 Nov 19. PMID 26585865
- [Background] Okoroha KR, Fidai MS, Tramer JS, Davis KD, Kolowich PA. Diagnostic accuracy of ultrasound for rotator cuff tears. Ultrasonography. 2019 Jul;38(3):215-220. doi: 10.14366/usg.18058. Epub 2018 Nov 17. PMID 30744304
- [Background] Okoroha KR, Mehran N, Duncan J, Washington T, Spiering T, Bey MJ, Van Holsbeeck M, Moutzouros V. Characterization of Rotator Cuff Tears: Ultrasound Versus Magnetic Resonance Imaging. Orthopedics. 2017 Jan 1;40(1):e124-e130. doi: 10.3928/01477447-20161013-04. Epub 2016 Oct 18. PMID 27755645
- [Background] Ostrander RV, Klauser JM, Menon S, Hackel JG. Ultrasound and Functional Assessment of Transtendinous Repairs of Partial-Thickness Articular-Sided Rotator Cuff Tears. Orthop J Sports Med. 2017 Mar 27;5(3):2325967117697375. doi: 10.1177/2325967117697375. eCollection 2017 Mar. PMID 28451606